CLINICAL TRIAL: NCT04103463
Title: Effects of Interactive Stepping Exercise on Memory in Adults With Amnestic Mild Cognitive Impairment
Brief Title: Interactive Stepping Exercise on Memory
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM108072F
Record Dates: First submitted 2019-09-20; First posted 2019-09-25 (Actual); Last update posted 2019-09-25 (Actual); Status verified 2019-09

CONDITIONS: Amnestic Mild Cognitive Impairment; Interactive Stepping Exercise; Memory; Cognitive Function; Executive Function
Keywords: square stepping exercise; Amnestic mild cognitive impairment; Interactive stepping exercise; memory; cognitive function; executive function

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interactive stepping exercise group (Experimental)
  Interventions: Other: Interactive stepping exercise
- Home exercise group (Active Comparator)
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Interactive stepping exercise — An exercise intervention based on the principle of square stepping exercise
  Arms: Interactive stepping exercise group
Other: Home exercise — Home exercise
  Arms: Home exercise group

SUMMARY:
This is a randomized controlled trail. A total of 28 individuals with aMCI will be randomly assigned to either the ISE group or control group. The ISE intervention conducts three times a week for 16 weeks. Outcomes are measured at baseline and after intervention. The primary outcomes are the Chinese version verbal learning test (CVVLT), selective reminding test (SRT), and logic memory test (Wechsler Memory Scale). The secondary outcomes are Montreal Cognitive Assessment (MoCA) for cognitive function, and trail making test Part A & B (TMT-A & B), Stroop test, and 25-item Executive Interview (C-EXIT 25) for executive function.

ELIGIBILITY:
Inclusion Criteria:

* Age≥50 years
* Complained of memory impairment
* Chinese Version Verbal Learning Test 10-minute delays ≤ 6 words
* MMSE score≥24 and CDR score=0.5
* Activities of daily living are intact
* DSM-IV criteria for the diagnosis of dementia is not met

Exclusion Criteria:

* Any significant neurologic disease other than suspected incipient Alzheimer's disease
* Psychotic features, contraindication of exercise... which could lead to difficulty complying with the protocol

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Chinese version verbal learning test | Change from baseline at 12 week
Selective reminding test | Change from baseline at 12 week
Wechsler Memory Scale-III | Change from baseline at 12 week
Logic memory test | Change from baseline at 12 week

SECONDARY OUTCOMES:
Montreal Cognitive Assessment | Change from baseline at 12 week
Trail making test | Change from baseline at 12 week
Stroop test | Change from baseline at 12 week
Executive Interview | Change from baseline at 12 week